CLINICAL TRIAL: NCT07174180
Title: The Effect of Wearing the Hijab on Dry and Evaporative Heat Exchange During Moderate-intensity Exercise Performed in Hot-dry Environments
Brief Title: The Impact of Wearing the Hijab on Whole-body Heat Loss During Exercise-heat Stress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Full Professor, University Research Chair, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HEPRU-2025-08-A
Record Dates: First submitted 2025-08-15; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Heat Stress; Temperature Change, Body
Keywords: Core temperature; Exercise; Females; Garment; Heat strain; Thermoregulation; Hot weather
MeSH Terms: conditions — Heat Stress Disorders; Body Temperature Changes; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No hijab (Experimental): Participants rest in a thermoneutral resting condition for 30-min (baseline resting) while wearing a cotton t-shirt and shorts, after which they enter a chamber regulated at 40°C where they perform an intermittent exercise bout consisting of two, 30-min moderate-intensity exercise bouts (fixed rate of heat production of 200 W/m2), with each exercise bout separated by a 15 min rest break and a 60-min recovery following the second exercise bout.
  Interventions: Other: Exercise-heat stress with no hijab
- Hijab (Experimental): Participants rest in a thermoneutral resting condition for 30-min (baseline resting) while wearing a hijab over cotton t-shir and shorts, after which they enter a chamber regulated at 40°C where they perform an intermittent exercise bout consisting of two, 30-min moderate-intensity exercise bouts (fixed rate of heat production of 200 W/m2), with each exercise bout separated by a 15 min rest break and a 60-min recovery following the second exercise bout.
  Interventions: Other: Exercise-heat stress with a hijab

INTERVENTIONS:
Other: Exercise-heat stress with no hijab — Participants perform exercise in the heat with no hijab
  Arms: No hijab
Other: Exercise-heat stress with a hijab — Participants perform exercise in the heat with a hijab
  Arms: Hijab

SUMMARY:
The hijab (headscarf and cloak) is a Muslim dress, which covers the head, neck and chest, and conceals the female hair, leaving the face uncovered. It is worn by Muslim women worldwide including young Muslim women engaging in sports and exercise. As with any clothing worn on the body, the hijab can impact heat dissipation during exercise, potentially leading to increased body temperature and discomfort, especially in warmer environments. However, the extent to which the hijab may restrict heat loss remains unclear. This study aims to assess dry and evaporative heat exchange in young women performing moderate-intensity intermittent exercise in dry heat conditions (40°C, 15% relative humidity).

ELIGIBILITY:
Inclusion Criteria:

* healthy young female (18-35 years)
* non smoking
* English or French speaking
* ability to provide informed consent

Exclusion Criteria:

* claustrophobia
* engaged in endurance training
* acute or chronic illness
* sedentary (not engaged in any form of physical activity)
* physical restriction limiting physical activity

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaporative heat loss at end exercise | End of the 60-min intermittent exercise bout
  Evaporative heat loss as assessed using a direct air calorimeter
Dry heat loss at end exercise | End of the 60-min intermittent exercise bout
  Dry heat loss as assessed using a direct air calorimeter
Total heat loss at end exercise | End of the 60-min intermittent exercise bout
  Total heat loss as assessed using a direct air calorimeter
Body heat storage | End of the 60-min intermittent exercise bout
  Heat stored in the body for each of the exercise bouts
Change in body heat content | End of the 60-min intermittent exercise bout
  Body heat content measured at the end of intermittent exercise
Core temperature | End of the 60-min intermittent exercise bout
  Rectal temperature during final 5 minutes of each of the exercise bouts
Mean skin temperature | End of the 60-min intermittent exercise bout
  Mean skin temperature during final 5 minutes of each of the exercise bouts
Relative change in core temperature at end exercise | End of the 60-min intermittent exercise bout
  Relative increase in core temperature for each 30-minute exercise bout
Relative change in mean skin temperature at end exercise | End of the 60-min intermittent exercise bout
  Relative change in mean skin temperature for each 30-minute exercise bout
Heart rate | End of the 60-min intermittent exercise bout
  Heart rate during final 5 minutes of each of the exercise bouts
Rating of perceived exertion | End of the 60-min intermittent exercise bout
  Perceived exertion assessed via a self-report questionnaire upon verbal prompting (scale is as follows: 6: indicating the participant is not exerting themselves at all with 20 indicating participant is exerting themselves maximally)
Thermal sensation A | End of the 60-min intermittent exercise bout
  Thermal sensation assessed via a self-report questionnaire upon verbal prompting (scale is as follows: 7-point scale; -3 indicating the participant is cold to +3 indicating the participant is hot)
Thermal sensation B | End of the 60-min intermittent exercise bout
  Thermal sensation assessed via a self-report questionnaire upon verbal prompting (scale is as follows: 7-point scale; 0 indicating the participant is neutral to 7 indicating the participant is extremely hot)
Thirst sensation | End of the 60-min intermittent exercise bout
  Thirst sensation assessed via a self-report questionnaire upon verbal prompting (scale is as follows: 9-point scale; 1 indicating the participant is not thirsty at all to 9 indicating the participant is very, very thirsty)

CONTACTS AND LOCATIONS:
Overall Officials: Glen P Kenny, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada